CLINICAL TRIAL: NCT05995054
Title: A Prospective, One-arm and Open Clinical Study to Assess Safety and Efficacy of Anti-Human CD20 Monoclonal Antibody Obinutuzumab in the Treatment of Primary Immune Thrombocytopenia
Brief Title: A Prospective, One-arm and Open Clinical Study of Obinutuzumab in the Treatment of Immune Thrombocytopenia
Acronym: 2023CD20ITP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023039
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-09

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Obinutuzumab) (Experimental): 110 enrolled subjects: one infusion
  Interventions: Drug: Obinutuzumab Injection [Gazyva]

INTERVENTIONS:
Drug: Obinutuzumab Injection [Gazyva] — intravenous Obinutuzumab administration
  This study adopts a prospective, single arm, open design method. 110 subjects were enrolled in the study and were treated with CD20 monoclonal antibody (Obinutuzumab: 1000mg) for once.
  The first stage is the main research stage (d1-w12), which is the core treatment period. The subjects will receive intravenous infusion of 1000mg Obinutuzumab for once to observe the safety and efficacy during treatment.
  The second stage (w12-w48) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy of Obinutuzumab after treatment.

SUMMARY:
To evaluate the safety and efficacy of Obinutuzumab in the treatment of immune thrombocytopenia in patients who have not responded adequately or relapsed after first-line treatment.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

Obinutuzumab is the first personalized type Ⅱ glycosylation engineered CD20 monoclonal antibody. Studies have shown that compared with rituximab, obinutuzumab may improve its efficacy in lymphoma by increasing DCD and ADCC effects and reducing drug resistance by reducing CDC effects. In view of this, Obinutuzumab may have the same effect in the treatment of ITP, and may be more effective in the treatment of ITP, but there is also a risk of poor efficacy. At present, there is a lack of data on the efficacy and safety of Obinutuzumab in the treatment of ITP in China.

Therefore, the investigators designed this clinical trial to evaluate the safety and efficacy of Obinutuzumab in the treatment of immune thrombocytopenia in patients who have not responded adequately or relapsed after first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female
* Conform to the diagnostic criteria of immune Thrombocytopenia (ITP)
* Diagnosis of ITP ≥3 months, and with a platelet count of <30 X 109/L measured within 2 days prior to administration（Platelet counts were measured at least 2 times during screening (at least 1 week apart) with platelets<30 X 109/L）
* Failure to achieve response or relapse after corticosteroid therapy
* The previous emergency treatment of ITP (e.g. methylprednisolone, platelet transfusion, IVIG transfusion) must be completed at least 2 weeks before the first administration
* Signed and dated written informed consent
* With Liver and kidney function<1.5×upper limit of normal， such as ALT、AST，BUN，Cre，etc.
* ECOG physical state score ≤ 2 points
* Cardiac function of the New York Society of Cardiac Function ≤ 2
* Patients receiving maintenance treatment (including corticosteroids (less than or equal to 0.5mg/kg prednisone), TPO receptor agonists, etc.) must have a stable dose at least 4 weeks before the first administration, and azathioprine, danazol, cyclosporin A, tacrolimus, sirolimus, etc. must be stopped at least 4 weeks before the first administration; The end of rituximab treatment was>3 months；More than 6 months after splenectomy.

Exclusion Criteria:

* Subjects with primary disease of important organs (liver, kidney, heart, etc.), or with immune system diseases;
* Secondary thrombocytopenia caused by various reasons, such as connective tissue disorders, bone marrow hematopoietic failure disease, myelodysplastic syndrome, malignancy, drugs, inherited thrombocytopenia, common variable immune deficiency, lymphoma, etc.;
* Subjects infected with human immunodeficiency virus (HIV);
* Uncontrollable or active infections during the screening period, including hepatitis B, hepatitis C, cytomegalovirus, EB virus, or positive syphilis antigen;
* Subjects with extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage;
* Subjects with heart disease that requires treatment or hypertension that has been judged by researchers to be poorly controlled currently;
* Subjects with any venous or arterial thrombosis, atherosclerosis, and other diseases;
* Subjects with a history of malignant solid tumor or have received allogeneic stem cell transplantation or organ transplantation;
* Subjects with mental disorders who are unable to sign normal informed consent and conduct trials and follow-up;
* Subjects whose toxic symptoms caused by pre-trial treatment have not disappeared;
* Subjects with other serious diseases that may limit their participation in this trial (diabetes; severe cardiac insufficiency; myocardial obstruction or unstable arrhythmia or unstable angina pectoris in the last 6 months; gastric ulcer; active autoimmune disease, etc.);
* Subjects with septicemia or other irregular bleeding;
* Female subjects who are nursing or pregnant/suspected pregnant (positive pregnancy tests for human chorionic gonadotropin in urine during screening).
* Patients taking antiplatelet drugs at the same time;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of overall efficacy response after Obinutuzumab treatment within 12 weeks | 12 weeks
  Overall response rate defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile within 12 weeks after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period

SECONDARY OUTCOMES:
Evaluation of overall efficacy response after Obinutuzumab treatment within 8 weeks | 8 weeks
  Overall response rate defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile within 8 weeks after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Evaluation of overall efficacy response after Obinutuzumab treatment within 6 months | 6 months
  Overall response rate defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile within 6 months after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Evaluation of overall efficacy response after Obinutuzumab treatment within 12 months | 12 months
  Overall response rate defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile within 12 months after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Evaluation of sustained response rate after Obinutuzumab treatment within 6 months | 6 months
  Sustained response rate defined as proportion of subjects who keep a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile at 6 months after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Evaluation of sustained response rate after Obinutuzumab treatment within 12 months | 12 months
  Sustained response rate defined as proportion of subjects who keep a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile at 12 months after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Time to onset response | 12 months
  Time to onset response defined as the time needed for subjects to have a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Duration of response | 12 months
  The longest duration for which the subject sustained a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline at the meanwhile after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Emergency treatment after Obinutuzumab treatment within 12 weeks | 12 weeks
  Percentage of subjects who received emergency treatment after Obinutuzumab treatment within 12 weeks
Reduction of concomitant drug after Obinutuzumab treatment within 12 weeks | 12 weeks
  Percentage of patients with reduced doses of corticosteroids and/or other concomitant immunosuppressive drugs at baseline by 12 weeks of Obinutuzumab treatment
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale after Obinutuzumab treatment within 12 weeks | 12 weeks
  Changes of the subjects' numbers in WHO bleeding score after Anti-CD20 antibody treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
One-year recurrence-free survival rate | 12 months
  Time from the start of treatment to the occurrence of a relapse or death event
Safety of Anti-CD20 antibody treatment | 12 months
  Incidence, severity, and relationship of treatment emergent adverse events after Anti-CD20 antibody treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI